CLINICAL TRIAL: NCT02514603
Title: A Phase 1 Study of LY2606368 in Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of Prexasertib (LY2606368) in Japanese Participants With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16018; I4D-JE-JTJK (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Neoplasm
Keywords: Neoplasm metastasis; Checkpoint Kinase 1; CHK1; CHK1 inhibitor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — prexasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prexasertib (Experimental): Prexasertib intravenously (IV) on day 1 of a 14 day cycle. Treatment with prexasertib may continue until disease progression, unacceptable toxicity, or other discontinuation criteria are met.
  Interventions: Drug: Prexasertib

INTERVENTIONS:
Drug: Prexasertib — Administered IV
  Other Names: LY2606368

SUMMARY:
The primary purpose of this study is to assess the tolerability of prexasertib in Japanese participants with advanced solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be appropriate candidate for experimental therapy, as determined by investigator, after available standard therapies have failed
* Participant must have diagnosis of cancer that is advanced or metastatic
* Participant must have discontinued previous treatments for cancer and recovered from the acute effects of that therapy
* If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for three months following the last dose of study drug
* If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 7 days of the first dose of study drug and must not be breast feeding

Exclusion Criteria:

* Participant must not have symptomatic central nervous system malignancy or metastasis
* Participant must not have current hematologic malignancy
* Participant must not have an active symptomatic fungal, bacterial or viral infection, including human immunodeficiency virus (HIV) or Hepatitis A, B, or C
* Participant must not have a serious cardiac condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Prexasertib Dose-Limiting Toxicities (DLT) | Cycle 1 (14 day cycle)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Prexasertib | Pre-dose up to 7 Days Post Treatment in Cycle 1/2 (Approximately 7 Days)
Pharmacokinetics (PK): Area Under Curve (AUC) of Prexasertib | Pre-dose up to 7 Days Post Treatment in Cycle1/2 (Approximately 7 Days)
Percentage of Participants with a Tumor Response | Baseline to Study Completion (Approximately 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo